CLINICAL TRIAL: NCT03466242
Title: IN Dexmedetomidine for Procedural Sedation in Pediatric Closed Reductions for Distal Forearm Fractures. Timmons Z MD, Feudale B MD Children Presenting to the ED With Distal Forearm Extremity Fractures Often Require Re-alignment Under Conscious Sedation. The Objective of This Study is to Evaluate the Sedative, and Analgesic Effects of Intranasal (IN) Dexmedetomidine (DEX) Who Undergo Conscious Sedation for Reduction of Closed Distal Forearm Fractures When Compared to Those Receiving the Standard of Care Intravenous (IV) Ketamine
Brief Title: IN Dexmedetomidine for Procedural Sedation in Pediatric Closed Reductions for Distal Forearm Fractures
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Never IRB reviewed or approved.
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-193
Record Dates: First submitted 2018-03-01; First posted 2018-03-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Conscious Sedation; Distal Radius Fracture
Keywords: intranasal dexmedetomidine
MeSH Terms: conditions — Wrist Fractures | interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Intervention Model Description: This will be a feasibility pilot study, and as such, will be non-blinded, and utilize a convenience sample of children aged 2-18 years old requiring closed reduction under conscious sedation for distal forearm fractures. 20 children recruited in IN Dex arm and 20 children in Ketamine arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal Dexmedetomidine (Experimental): Evaluate sedative and analgesic effects of Intranasal Dexmedetomidine (1-2ug/kg)
  Interventions: Drug: Dexmedetomidine
- IV Ketamine (Active Comparator): Evaluate sedative and analgesic effects of Intravenous Ketamine (1mg/kg)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — Evaluate sedative and analgesic effects of Intranasal Dexmedetomidine
  Other Names: Precedex
  Arms: Intranasal Dexmedetomidine
Drug: Ketamine — Evaluate sedative and analgesic effects of Intravenous Ketamine
  Arms: IV Ketamine

SUMMARY:
The primary objective of this study is to evaluate the sedative, and analgesic effects of intranasal (IN) Dexmedetomidine (DEX) in children presenting to a Pediatric Emergency Department (PED) who undergo conscious sedation for reduction of closed distal forearm fractures when compared to those receiving intravenous (IV) Ketamine. The secondary objective is to compare each sedation technique for safety and procedural outcomes.

DETAILED DESCRIPTION:
Distal Forearm fractures are often are displaced requiring conscious sedation for closed reduction in the Emergency Department. Our institution's current standard of care consists of IN Fentanyl for baseline control of pain, and for those fractures requiring reduction; typically IV Ketamine is utilized. Ketamine is typically well tolerated but is not without concerns including hypertension, vomiting, and the rare but serious complication of laryngospasm. Dexmedetomidine (DEX) offers a possible alternative to IV Ketamine. DEX has been used safely in the critical care setting for both pediatrics and adults. It has been well documented as being quite effective in sedation, amnesia and analgesia. Using IN DEX for PED procedural sedation has the potential to obviate the need for IV placement and may offer a better conscious sedation profile than Ketamine with respect to sedation, analgesia, and adverse outcomes.

Our overall project would be to assess the efficiency of IN DEX in comparison to IV Ketamine, for proper sedation and analgesic coverage for children undergoing closed reduction of distal forearm fractures.

ELIGIBILITY:
Inclusion Criteria:Verbal children aged 2-18 with a single extremity displaced forearm fracture requiring conscious sedation and reduction will be screened for enrollment.

Exclusion Criteria:

1. Under age 2 years old or patients > 18 years old
2. Multiple Fractures
3. Significant multisystem trauma
4. Glasgow Coma Scale (GCS < 15)
5. Complex fractures that aren't deemed reducible in ED
6. Reported Allergy to Alpha -2-agonists
7. Pregnancy
8. Intoxication
9. Baseline Hypotension as < 70mm Hg + 2 x age or < 90mm Hg for patients > 11 years of age
10. Patients with prior reductions attempted at outside facilities
11. Aberrant nasal anatomy that precludes IN medications
12. Chronic Health issues that can affect DEX metabolism
13. History of adverse reactions to anesthesia
14. Patients transferred from outside facilities
15. Open fractures

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sedative effects of intranasal Dexmedetomidine in children undergoing conscious sedation for closed distal forearm fracture reduction compared to intravenous Ketamine | 12 months
  The sedative effects of intranasal Dexmedetomidine will be compared to intravenous ketamine for conscious sedation via the Michigan Sedation Scoring (MSS) system.
Evaluate the analgesic effects of intranasal Dexmedetomidine in children undergoing conscious sedation for closed distal forearm fracture reduction compared to intravenous Ketamine | 12 months
  The analgesic effects of intranasal Dexmedetomidine will be compared to intravenous ketamine for conscious sedation using either the Wong-Baker scale (FACES) or Visual Analogue Scale (VAS) depending on patient age and developmental status

SECONDARY OUTCOMES:
Compare each sedation technique for time to sedation onset | 12 months
  Time in minutes and seconds from administration of sedative agent until Michigan Sedation Scoring (MSS) is 3 or higher.
Compare each sedation technique for length of sedation | 12 months
  Time in minutes and seconds from when Michigan Sedation Scoring (MSS) is 3 or higher until MSS is less than 3.
Compare each sedation technique for length of ED stay | 12 months
  Time in minutes and seconds from presentation to ED to discharge
Compare each sedation technique for need for additional doses of medications for analgesia or sedation | 12 months
  Will measure if any unplanned doses of sedatives or analgesics are required in either treatment arm.
Compare each sedation technique for Vital sign abnormalities | 12 months
  Review vital signs following administration of either study drug to see if any vital signs were abnormal. Abnormal vital signs will be defined as hear rate, respiratory rate, or blood pressure above or below one standard deviation for age derived norms.
Compare each sedation technique for need for respiratory interventions | 12 months
  Measure if any respiratory interventions were required during the patient's ED stay. Respiratory interventions defined as need for oxygen by any device.
Compare each sedation technique for rate of vomiting | 12 months
  Describe the incidence (yes/no) of vomiting at any point after administration of either study drug to ED discharge.
Compare each sedation technique for procedural success rate | 12 months
  Describe the successful reduction of orthopedic injuries in each study arm. Successful reduction defined as patient able to be discharged and not requiring admission, surgery, or secondary reduction attempts.
Compare each sedation technique for patient family satisfaction | 12 months
  Describe the family satisfaction with each conscious sedation technique. Measured by brief survey given to the family upon consent for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zebulon Timmons, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Landin LA. Epidemiology of children's fractures. J Pediatr Orthop B. 1997 Apr;6(2):79-83. doi: 10.1097/01202412-199704000-00002. PMID 9165435
- [Result] Gausche-Hill M, Brown KM, Oliver ZJ, Sasson C, Dayan PS, Eschmann NM, Weik TS, Lawner BJ, Sahni R, Falck-Ytter Y, Wright JL, Todd K, Lang ES. An Evidence-based Guideline for prehospital analgesia in trauma. Prehosp Emerg Care. 2014;18 Suppl 1:25-34. doi: 10.3109/10903127.2013.844873. Epub 2013 Nov 26. PMID 24279813
- [Result] Borland M, Jacobs I, King B, O'Brien D. A randomized controlled trial comparing intranasal fentanyl to intravenous morphine for managing acute pain in children in the emergency department. Ann Emerg Med. 2007 Mar;49(3):335-40. doi: 10.1016/j.annemergmed.2006.06.016. Epub 2006 Oct 25. PMID 17067720
- [Result] Litke J, Pikulska A, Wegner T. Management of perioperative stress in children and parents. Part I--the preoperative period. Anaesthesiol Intensive Ther. 2012 Jul-Sep;44(3):165-9. PMID 23110295
- [Result] Bhat R, Santhosh MC, Annigeri VM, Rao RP. Comparison of intranasal dexmedetomidine and dexmedetomidine-ketamine for premedication in pediatrics patients: A randomized double-blind study. Anesth Essays Res. 2016 May-Aug;10(2):349-55. doi: 10.4103/0259-1162.172340. PMID 27212773
- [Result] Miller K, Tan X, Hobson AD, Khan A, Ziviani J, O'Brien E, Barua K, McBride CA, Kimble RM. A Prospective Randomized Controlled Trial of Nonpharmacological Pain Management During Intravenous Cannulation in a Pediatric Emergency Department. Pediatr Emerg Care. 2016 Jul;32(7):444-51. doi: 10.1097/PEC.0000000000000778. PMID 27380603
- [Result] Fowler-Kerry S, Lander JR. Management of injection pain in children. Pain. 1987 Aug;30(2):169-175. doi: 10.1016/0304-3959(87)91072-4. PMID 3670868
- [Result] Kogan A, Katz J, Efrat R, Eidelman LA. Premedication with midazolam in young children: a comparison of four routes of administration. Paediatr Anaesth. 2002 Oct;12(8):685-9. doi: 10.1046/j.1460-9592.2002.00918.x. PMID 12472704
- [Result] Iirola T, Vilo S, Manner T, Aantaa R, Lahtinen M, Scheinin M, Olkkola KT. Bioavailability of dexmedetomidine after intranasal administration. Eur J Clin Pharmacol. 2011 Aug;67(8):825-31. doi: 10.1007/s00228-011-1002-y. Epub 2011 Feb 12. PMID 21318594
- [Result] Phan H, Nahata MC. Clinical uses of dexmedetomidine in pediatric patients. Paediatr Drugs. 2008;10(1):49-69. doi: 10.2165/00148581-200810010-00006. PMID 18162008
- [Result] Behrle N, Birisci E, Anderson J, Schroeder S, Dalabih A. Intranasal Dexmedetomidine as a Sedative for Pediatric Procedural Sedation. J Pediatr Pharmacol Ther. 2017 Jan-Feb;22(1):4-8. doi: 10.5863/1551-6776-22.1.4. PMID 28337075
- [Result] Yuen VM, Hui TW, Irwin MG, Yao TJ, Wong GL, Yuen MK. Optimal timing for the administration of intranasal dexmedetomidine for premedication in children. Anaesthesia. 2010 Sep;65(9):922-9. doi: 10.1111/j.1365-2044.2010.06453.x. PMID 20645951
- [Result] Yuen VM, Hui TW, Irwin MG, Yao TJ, Chan L, Wong GL, Shahnaz Hasan M, Shariffuddin II. A randomised comparison of two intranasal dexmedetomidine doses for premedication in children. Anaesthesia. 2012 Nov;67(11):1210-6. doi: 10.1111/j.1365-2044.2012.07309.x. Epub 2012 Sep 5. PMID 22950484
- [Result] Miller JW, Divanovic AA, Hossain MM, Mahmoud MA, Loepke AW. Dosing and efficacy of intranasal dexmedetomidine sedation for pediatric transthoracic echocardiography: a retrospective study. Can J Anaesth. 2016 Jul;63(7):834-41. doi: 10.1007/s12630-016-0617-y. Epub 2016 Feb 16. PMID 26883963
- [Result] Reynolds J, Rogers A, Capehart S, Manyang P, Watcha MF. Retrospective Comparison of Intranasal Dexmedetomidine and Oral Chloral Hydrate for Sedated Auditory Brainstem Response Exams. Hosp Pediatr. 2016 Mar;6(3):166-71. doi: 10.1542/hpeds.2015-0152. PMID 26917547
- [Result] Malhotra PU, Thakur S, Singhal P, Chauhan D, Jayam C, Sood R, Malhotra Y. Comparative evaluation of dexmedetomidine and midazolam-ketamine combination as sedative agents in pediatric dentistry: A double-blinded randomized controlled trial. Contemp Clin Dent. 2016 Apr-Jun;7(2):186-92. doi: 10.4103/0976-237X.183058. PMID 27307665
- [Result] Li BL, Zhang N, Huang JX, Qiu QQ, Tian H, Ni J, Song XR, Yuen VM, Irwin MG. A comparison of intranasal dexmedetomidine for sedation in children administered either by atomiser or by drops. Anaesthesia. 2016 May;71(5):522-8. doi: 10.1111/anae.13407. Epub 2016 Mar 3. PMID 26936022
- [Result] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Result] Ebert TJ, Hall JE, Barney JA, Uhrich TD, Colinco MD. The effects of increasing plasma concentrations of dexmedetomidine in humans. Anesthesiology. 2000 Aug;93(2):382-94. doi: 10.1097/00000542-200008000-00016. PMID 10910487
- [Result] Olutoye O, Kim T, Giannoni C, Stayer S. Dexmedetomidine as an analgesic for pediatric tonsillectomy and adenoidectomy. Paediatr Anaesth. 2007 Oct;17(10):1007-8. doi: 10.1111/j.1460-9592.2007.02234.x. No abstract available. PMID 17767643
- [Result] Sheta SA, Al-Sarheed MA, Abdelhalim AA. Intranasal dexmedetomidine vs midazolam for premedication in children undergoing complete dental rehabilitation: a double-blinded randomized controlled trial. Paediatr Anaesth. 2014 Feb;24(2):181-9. doi: 10.1111/pan.12287. Epub 2013 Nov 15. PMID 24237879
- [Result] Niesters M, Martini C, Dahan A. Ketamine for chronic pain: risks and benefits. Br J Clin Pharmacol. 2014 Feb;77(2):357-67. doi: 10.1111/bcp.12094. PMID 23432384
- [Result] Lightdale JR, Mitchell PD, Fredette ME, Mahoney LB, Zgleszewski SE, Scharff L, Fox VL. A Pilot Study of Ketamine versus Midazolam/Fentanyl Sedation in Children Undergoing GI Endoscopy. Int J Pediatr. 2011;2011:623710. doi: 10.1155/2011/623710. Epub 2011 May 16. PMID 21760813
- [Result] Rasmussen KG. Psychiatric side effects of ketamine in hospitalized medical patients administered subanesthetic doses for pain control. Acta Neuropsychiatr. 2014 Aug;26(4):230-3. doi: 10.1017/neu.2013.61. PMID 25142291
- [Result] Parvizrad R, Pakniyat A, Malekianzadeh B, Almasi-Hashiani A. Comparing the analgesic effect of intranasal with intravenous ketamine in isolated orthopedic trauma: A randomized clinical trial. Turk J Emerg Med. 2017 Jun 23;17(3):99-103. doi: 10.1016/j.tjem.2017.05.006. eCollection 2017 Sep. PMID 28971157
- [Result] Jonkman K, Dahan A, van de Donk T, Aarts L, Niesters M, van Velzen M. Ketamine for pain. F1000Res. 2017 Sep 20;6:F1000 Faculty Rev-1711. doi: 10.12688/f1000research.11372.1. eCollection 2017. PMID 28979762